CLINICAL TRIAL: NCT00020397
Title: Immunization Of HLA-A*0201 or HLA-DPB1*04 Patients With Metastatic Melanoma Using Epitopes From The ESO-1 Antigen
Brief Title: Vaccine Therapy in Treating Patients With Refractory Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068403; NCI-01-C-0032; NCI-2390; NCT00006491 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2005-01

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

INTERVENTIONS:
Biological: NY-ESO-1 peptide vaccine
Biological: aldesleukin

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of vaccine therapy in treating patients who have refractory metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether an immunologic response can be obtained after administration of ESO-1 peptide vaccine comprising class I , II, or both peptides in HLA-A*201 or HLA-DPB1*04 positive patients with refractory metastatic melanoma expressing ESO-1.
* Determine the toxicity of this vaccine in these patients.
* Determine whether prior immunization with this vaccine results in increased clinical responsiveness in patients treated with interleukin-2.

OUTLINE: Patients are assigned to 1 of 3 groups according to HLA type.

* Group 1 (HLA-A*201 and HLA-DPB1*04 positive): Patients receive ESO-1 peptide vaccine comprising class I (ESO-1:157-165 [165V]) and class II (ESO-1:161-180) peptides subcutaneously once every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
* Group 2 (HLA-A*201 positive and HLA-DPB1*04 negative):Patients receive ESO-1 peptide vaccine as in group I comprising class I peptide only.
* Group 3 (HLA-A*201 negative and HLA-DPB1*04 positive):Patients receive ESO-1 peptide vaccine as in group I comprising class II peptide only.

Patients who develop disease progression discontinue vaccinations and receive high-dose interleukin (IL-2) IV over 15 minutes every 8 hours for up to 4 days (maximum of 12 doses). Treatment with IL-2 repeats every 10-14 days for 4 courses in the absence of disease progression (after at least 2 courses) or unacceptable toxicity.

Patients who have stable disease or a mixed or partial response to vaccination or IL-2 therapy may be eligible for additional vaccine therapy. Patients who have a complete response to vaccine therapy are eligible for 1 additional treatment.

Patients are followed at 3 weeks.

PROJECTED ACCRUAL: A total of 45-90 patients (15-30 per treatment group) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma that expresses ESO-1 antigen
* Must have progressed during prior standard treatment
* Measurable or evaluable disease
* HLA-A*201 or HLA-DPB1*04 positive

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 90,000/mm^3

Hepatic:

* SGOT and SGPT less than 3 times normal
* Bilirubin no greater than 1.6 mg/dL (3.0 mg/dL for patients with Gilbert's syndrome)
* Hepatitis B surface antigen negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No cardiac ischemia*
* No myocardial infarction*
* No cardiac arrhythmias* NOTE: *For interleukin-2 (IL-2) administration

Pulmonary:

* No obstructive or restrictive pulmonary disease (for IL-2 administration)

Immunologic:

* No autoimmune disease
* No active primary or secondary immunodeficiency
* HIV negative
* No active systemic infections

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active major medical illness (for IL-2 administration)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior ESO-1 immunization

Chemotherapy:

* Recovered from any prior chemotherapy

Endocrine therapy:

* No concurrent systemic steroid therapy

Radiotherapy:

* Recovered from any prior radiotherapy

Surgery:

* Not specified

Other:

* At least 3 weeks since any prior systemic therapy for cancer
* No other concurrent systemic therapy for cancer

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-11; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Khong HT, Yang JC, Topalian SL, Sherry RM, Mavroukakis SA, White DE, Rosenberg SA. Immunization of HLA-A*0201 and/or HLA-DPbeta1*04 patients with metastatic melanoma using epitopes from the NY-ESO-1 antigen. J Immunother. 2004 Nov-Dec;27(6):472-7. doi: 10.1097/00002371-200411000-00007. PMID 15534491